CLINICAL TRIAL: NCT04224909
Title: Video HIT Results in Sudden Sensorineural Hearing Loss Patients
Brief Title: Video HIT in Sudden Sensorineural Hearing Loss
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0633-19-TLV
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Sudden Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sudden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with Sudden Sensorineural Hearing Loss
  Interventions: Diagnostic Test: Video Head Impulse Test

INTERVENTIONS:
Diagnostic Test: Video Head Impulse Test — Diagnosis of dysfunction of the semicircular canals using the vHIT

SUMMARY:
The function of the vestibular system among patients with Sudden Sensori Neural Hearing Loss will be evaluted using the video Head Impulse Test

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with the diagnosis of Sudden Sensorineural Hearing Loss

Exclusion Criteria:

* Vertigo
* Other etiology causing dizziness
* Neurological dysfunction othe than the hearing loss
* Difficulty performing the vHIT
* Chronic vestibular disorder
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Sudden Sensorineural Hearing Loss
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
The gain of each canal, as calculated using the vHIT | 15 minutes
  Gain measured by the vHIT system

IPD SHARING:
Plan to Share IPD: No